CLINICAL TRIAL: NCT02346812
Title: Brassica Intake and Isothiocyanate Absorption: Intake Patterns May Have Implications for Cancer Prevention by Dietary Brassica Vegetables
Brief Title: Brassica Intake and Isothiocyanate Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HS49
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brassica (Experimental): Brassica vegetables will be consumed daily as part of a controlled diet.
  Interventions: Other: Controlled diet with brassica vegetables
- Control (Other): Typical American diet will be consumed, without any Brassica vegetables.
  Interventions: Other: Controlled diet without brassica vegetables

INTERVENTIONS:
Other: Controlled diet without brassica vegetables — Participants will be fed a controlled diet containing foods of a typical American diet.
  Arms: Control
Other: Controlled diet with brassica vegetables — Participants will be fed a controlled diet containing foods of a typical American diet.
  Arms: Brassica

SUMMARY:
Healthy individuals (n=18) will participate in 2 controlled-feeding study periods that are 3 weeks each in length: 1) Control diet 2) Brassica diet. The control diet will consist of typical American foods and will be free of Brassica vegetables and free of glucosinolates and isothiocyanates. The Brassica diet will contain the control diet plus glucosinolate/isothiocyanate treatment foods. There will be a break of 3 weeks in between study periods. Blood, urine, and fecal samples will be collected at the end of each study period. Eligible participants will be selected based on genotype for glutathione S-transferase (GST), which has been shown to influence the potential protective role of dietary Brassicas. Half the participants (n=9) will be GSTM1-positive individuals and half (n=9) will have the GSTM1-null genotype.

ELIGIBILITY:
Inclusion Criteria:

* Between 21 - 70 years of age
* Not currently taking glucosinolate/ITC containing supplements
* Voluntarily agree to participate and sign an informed consent document
* Free of cancer (never diagnosed or cancer-free for at least 5 y)

Exclusion Criteria:

* Pregnant, lactating, or intend to become pregnant during the study period
* Known allergy or intolerance to Brassica vegetables
* History of bariatric surgery or nutrient malabsorption disease (such as celiac disease) or other metabolic disorders requiring special diet recommendations
* Use of tobacco products
* Use of certain medications (prescription or over-the-counter) that may interfere with the study objectives
* Type 2 diabetes requiring the use of diabetes pills, insulin, or non-insulin shots
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol, or Miradon (anisindione)
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Total isothiocyanates (ITC) | 24-hr
  At the end of each study period, total ITC equivalents will be measured in blood and urine over a 24-hour period.

SECONDARY OUTCOMES:
Fecal microbiota | End of 3-week study period
  Fecal microbiota will be measured at the end of each 3-week study period.
Gastrointestinal health | 8-hr
  At the end of each 3-week study period, urine will be collected for 8 hours as part of the lactulose-mannitol test, which is a measure of gastrointestinal health.

CONTACTS AND LOCATIONS:
Locations (1):
- US Department of Agriculture Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Charron CS, Vinyard BT, Ross SA, Seifried HE, Jeffery EH, Novotny JA. Absorption and metabolism of isothiocyanates formed from broccoli glucosinolates: effects of BMI and daily consumption in a randomised clinical trial. Br J Nutr. 2018 Dec;120(12):1370-1379. doi: 10.1017/S0007114518002921. PMID 30499426